CLINICAL TRIAL: NCT04875156
Title: The Angle of the Metacarpophalangeal Joint of the Thumb During Maximal Pinch Strength: Implications for Arthrodesis
Brief Title: The Angle of the Metacarpophalangeal Joint of the Thumb During Maximal Pinch Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-08063
Record Dates: First submitted 2021-04-13; First posted 2021-05-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Post-traumatic; Arthrosis; Osteoarthritis Thumb
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: measurement of the joint mobility and the force of the thumb
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- normal volunteers (Other): normal volunteers between 18 and 40 years old, men and women. Measurement of the range of motion of the metacarpophalangeal joint with a goniometer and pinch strength of the thumb with a dynamometer
  Interventions: Other: measurement of range of motion and strength

INTERVENTIONS:
Other: measurement of range of motion and strength — measurement of range of motion (goniometer) and strength (dynamometer) of the metacarpophalangeal joint of the thumb

SUMMARY:
The aim of the study is to measure the position of the metacarpophalangeal joint of the thumb during key-pinch, tripod-pinch and opposition-pinch in normal volunteers, to determine the optimal position of metacarpophalangeal joint arthrodesis.

DETAILED DESCRIPTION:
The aim of the study is to measure the position of the metacarpophalangeal (MCP) joint of the thumb during key-pinch, tripod-pinch and opposition-pinch in normal volunteers, to determine the optimal position of metacarpophalangeal joint arthrodesis.

The force will be measured in three positions (key-pinch, tripod-pinch and opposition-pinch). Also measured is the degree of flexion of the MCP joint of the thumb. The mobility of the MCP joint of the thumb in maximum flexion and extension will also be measured. A total of about 300 healthy volunteers will be examined, with no history of trauma or disease to tendons or joints of the thumbs and between the ages of 18 and 40. The sponsor of this study is Professor Nadine Hollevoet. Master students of medicine from the faculty of medicine and health sciences will be part of the research team.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years

Exclusion Criteria:

* (previous) pathology of the joints, ligaments or tendons of the thumb

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
pinch strength of the thumb (in kilograms force) | 10 minutes
  pinch strength of the thumb in key-pinch, opposition-pinch and tripod-pinch
the angle of the metacarpophalangeal joint of the thumb (in degrees) | 10 minutes
  the angle of the metacarpophalangeal joint of the thumb (in degrees) during maximal force in the three pinch positions
range of motion of the metacarpophalangeal joint of the thumb (in degrees) | 10 minutes
  range of motion of the metacarpophalangeal joint of the thumb (in degrees) measuring maximal flexion and maximal extension of the joint

CONTACTS AND LOCATIONS:
Overall Officials: Nadine I Hollevoet, Phd, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gryson T, Van Der Velde G, Hollevoet N. Metacarpophalangeal joint angle of the thumb during maximal pinch strength: a study of healthy volunteers. J Hand Surg Eur Vol. 2023 Dec;48(11):1229-1230. doi: 10.1177/17531934231184821. Epub 2023 Jul 3. PMID 37401127